CLINICAL TRIAL: NCT05080010
Title: Three Cycles of Adjuvant Chemotherapy for the Patients With High-risk Retinoblastoma After Enucleation: Prospective Study
Brief Title: Adjuvant Chemotherapy for High-risk Postenucleation Retinoblastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Sun Yat-sen University, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yanghs2020
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Vincristine; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 cycles chemotherapy (Experimental): Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first three months.
  Interventions: Drug: 3 cycles chemotherapy

INTERVENTIONS:
Drug: 3 cycles chemotherapy — Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first three months.
  Other Names: vincristine, carboplatin, etoposide

SUMMARY:
The purpose of this study is to determine the effect of 3 cycles of chemotherapy(CEV) in the treatment of Stage I enucleated retinoblastoma.

DETAILED DESCRIPTION:
This study will be a phase Ⅲ open label interventional case series. Patients with Stage I enucleated retinoblastoma will receive 3 cycles of chemotherapy(CEV) oon a monthly basis. Patients will be followed for 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Definite pathology signs of retinoblastoma, Stage I base on International Retinoblastoma Staging System.
* Received enucleation in the study eye.
* Monocular retinoblastoma.

Exclusion Criteria:

* Any previous disease in the study eye.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals).
* History of chemical intervention for retinoblastoma in the study eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | five years
  measure the disease-free survival rate at five years

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, M.D, PHD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No